CLINICAL TRIAL: NCT01264887
Title: Open-label, Single-arm, Flexible Dosing, Phase III Trial, With Oral Tapentadol Prolonged Release (PR) in Subjects With Chronic Malignant Tumor-related Pain Who Have Completed the Maintenance Period of the KF5503/15 Trial.
Brief Title: Tapentadol in Chronic Malignant Tumour Related Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF5503/52; 2009-013291-46 (EudraCT Number); 168935 (Other: Grünenthal GmbH)
Record Dates: First submitted 2010-12-16; First posted 2010-12-22 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Cancer; Chronic Pain; Pain
Keywords: analgesia; analgesics; chronic pain; tumour related pain; chronic malignant tumor-related pain
MeSH Terms: conditions — Neoplasms; Chronic Pain; Pain; Agnosia | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tapentadol Prolonged Release (Experimental): Participants allocated to this treatment arm can be flexibly dosed between 100 to 250 mg tapentadol twice daily (50 and 100 mg tablets to be dispensed).
  Interventions: Drug: Tapentadol Prolonged Release

INTERVENTIONS:
Drug: Tapentadol Prolonged Release — Titration to achieve sufficient pain relief to continue with effective analgesia for as long as the participant tolerates and wishes to continue treatment.
  Other Names: Nucynta®; Palexia®; Yantil®

SUMMARY:
The purpose of this trial is the characterization of the long term safety profile and long-term dose requirements of tapentadol PR (prolonged release) in patients with malignant tumor-related pain. In the United States the prolonged-release formulation is also referred to as the extended-release formulation.

DETAILED DESCRIPTION:
The prevalence of tumor-related pain is high and the treatment of chronic tumor-related pain remains a challenging therapeutic problem.

Participants directly entering the KF5503/52 trial from the KF5503/15 trial (i.e., within 7 days of Visit 8 of the KF5503/15 trial) is scheduled: a Transfer Visit, an Open-label Treatment Period and a Follow-up Period.

For participants with a gap of more than 7 days and less than 24 weeks, between their full completion of the KF5503/15 trial and entry into the KF5503/52 trial the following is scheduled: an Enrollment Visit, an Entry Visit for assessment of eligibility, an Open-label Treatment Period and a Follow-up Period.

This trial was designed to offer patients with chronic malignant tumor-related pain the option of continuing treatment by receiving tapentadol prolonged release (PR).

The protocol scheduled visits every 28 days during the open-label treatment period. Unscheduled visits (or at least unscheduled telephone calls) were planned when dose adjustment is required. If a visit is not possible at the time of dose change, it could be done up to 7 days later. Unscheduled visits could also be performed whenever considered necessary (i.e., for evaluation of adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed an Informed Consent Form.
* At least 18 years of age.
* Male and non-pregnant, non-lactating female subjects. Sexually active women must be post menopausal, surgically sterile, or practicing an effective method of birth control before entry and throughout the trial. Female participants of child-bearing potential must have a negative pregnancy test at enrollment.
* Within 24 weeks of either full completion or completion of the double-blind treatment period (Visit 8) of KF5503/15 trial performed in participants with moderate to severe chronic malignant tumor related pain.
* Participant is, in the opinion of the investigator, expected to continue to have an overall positive benefit/risk ratio from continuing analgesic treatment within this trial.
* Participant must be willing to take tapentadol prolonged release (PR) throughout their participation in the trial.

Exclusion Criteria:

* History of alcohol and/or drug abuse.
* The participant has a clinically significant disease other than cancer that in the Investigator's opinion may affect the safety of the participant.
* Employees of the investigator or trial center or family members of the employees or the investigator.
* Known to or suspected of not being able to comply with the protocol and the use of tapentadol prolonged release (PR).
* Concurrent participation in another trial (except for participation in the KF5503/15 trial) or planning to be enrolled in another clinical trial during the course of this trial.
* Previous participation in another trial between the end of KF5503/15 and enrollment into the current trial, KF5503/52.
* History of seizure disorder, epilepsy, traumatic brain injury, stroke or transient ischemic attack.
* Known history and/or presence of cerebral tumors or metastases.
* Rapidly escalating pain or pain uncontrolled by therapy and was previously treated with maximum dose level of Investigational Medicinal Product.
* Participant is taking any prohibited concomitant medications.
* Uncontrolled hypertension.
* Known moderate or severe hepatic impairment.
* Known severe renal impairment.
* Clinically relevant history of hypersensitivity, allergy, or contraindications to tapentadol or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Georg Kress, Prof. Dr. med, Principal Investigator — General Hospital Vienna
Locations (12):
- Site 359004, Shumen, Bulgaria
- Hungary (2):
  - Site 036002, Nyíregyháza
  - Site 036010, Szekszárd
- Site 373001, Chisinau, Moldova
- Poland (2):
  - Site 048004, Bydgoszcz
  - Site 048001, Warsaw
- Romania (2):
  - Site 040006, Brasov
  - Site 040002, Bucharest
- Russia (2):
  - Site 007007, Nizhny Novgorod
  - Site 007012, Vladikavkaz
- Serbia (2):
  - Site 381001, Kamenitz
  - Site 381002, Niš

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on the 03 March 2011 and the last participant completed the trial on the 08 May 2014.
Groups:
- Tapentadol Prolonged Release: All participants from the KF5503/15 that enrolled into this trial were on tapentadol prolonged release. Participants were dosed in the range of 100 to 250 mg tapentadol twice daily. The dose was titrated to achieve sufficient pain relief to continue with effective analgesia for as long as the participant tolerated and wishes to continue treatment.
Period: Overall Study
Arm/Group | Tapentadol Prolonged Release
Started | 31
Completed | 0
Not Completed | 31
Not completed — Adverse Event | 5
Not completed — Death | 7
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 6
Not completed — Sponsor Decision Administrative Reasons | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Serbia | 6
  Hungary | 4
  Poland | 5
  Romania | 5
  Russian Federation | 3
  Bulgaria | 2
  Moldova, Republic of | 6
Weight [Mean (Standard Deviation); unit: kilograms] | 64.6 (16.45)
Height [Mean (Standard Deviation); unit: centimeters] | 165.0 (10.24)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (4.79)
Pain type [Number; unit: participants] — A participant could be suffering from more than one type of pain. The participant was counted in more than one category and therefore the addition of numbers are higher than the number of participants.
  participants
    Neuropathic | 23
    Visceral | 22
    Nociceptive (somatic) | 26

OUTCOME MEASURES:

1. Primary Outcome: Severity of Adverse Events
Description: The severity of treatment emergent adverse events was any untoward medical occurrence in a patient administered tapentadol. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of the (investigational) medicinal product whether or not related to the use of tapentadol.
  The clinical "intensity" of adverse event were classified as:
  Mild: signs and symptoms which can be easily tolerated. Symptoms could be ignored and disappeared when the participant is distracted.
  Moderate: symptoms caused discomfort but were tolerable, they could not be ignored and affect concentration.
  Severe: symptoms affected the usual daily activity.
Time Frame: Day 1; up to 144 weeks
Population: Safety Set.
Measure: Number; unit: participants
Groups:
- Number of Treatment Emergent Adverse Events: All participants from the KF5503/15 that enrolled into this trial were on tapentadol prolonged release. Participants were dosed in the range of 100 to 250 mg tapentadol twice daily. The dose was titrated to achieve sufficient pain relief to continue with effective analgesia for as long as the participant tolerated and wishes to continue treatment.
Arm/Group | Number of Treatment Emergent Adverse Events
Number analyzed (Participants) | 31
participants
  mild intensity | 3
  moderate intensity | 15
  severe intensity | 12

2. Secondary Outcome: Assess Consumption of Tapentadol During Long Term Use
Description: Summary of the modal total daily dose during the treatment period. The modal dose was based on assessment of the consecutive morning and evening intake amounts on each day and evaluation of the total daily dose.
Time Frame: Day 1; up to 144 weeks
Population: The modal dose is based on assessment of the consecutive morning and evening intake amounts on each day and evaluation of the total daily dose.
  No participant received more than 500 mg per day.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
participants
  less than 200 mg/day | 0
  200 to less than 250 mg/day | 3
  250 to less than 300 mg/day | 1
  300 to less than 350 mg/day | 8
  350 to less than 400 mg/day | 0
  400 to less than 450 mg/day | 11
  450 to less than 500 mg/day | 0
  500 mg/day | 8

3. Primary Outcome: Relatedness Assessment of Treatment Emergent Adverse Events
Description: Participant-based analysis of treatment emergent adverse events (TEAEs) regarding the relationship to the study drug (tapentadol). The TEAEs were reported by the participants or were captured by the investigator. The relationship was rated by the investigator. The categorization of relatedness into one of the two categories was based on the following: Related included "possible", "probable/likely", and "certain"; whilst unrelated treatment emergent adverse events include those rated by the investigator as "unlikely", "conditional/unclassified", "un-assessable/unclassifiable", and "not related".
Time Frame: Day 1; up to 144 weeks
Population: Safety Set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
participants
  No Treatment Emergent Adverse Events | 1
  All Treatment Emergent Adverse Events | 30
  Investigator-rated Related | 6
  Investigator-rated Not Related | 24

4. Primary Outcome: Countermeasures Taken Due to Treatment Emergent Adverse Events
Description: Participant-based analysis of treatment emergent adverse events (TEAEs) regarding countermeasure to the study drug (tapentadol). The TEAEs were reported by the participants or were captured by the investigator. The countermeasure taken by the investigator were reported.
Time Frame: Day 1; up to 144 weeks
Population: Safety Set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
participants
  All Treatment Emergent Events | 30
  No Treatment Emergent Adverse Events | 1
  No countermeasures taken | 5
  Countermeasures with Medication | 17
  Trial Discontinued Countermeasure | 6
  Other Countermeasure due to Somnolence | 1
  Other Countermeasure due to Migraine | 1

5. Other Pre Specified Outcome: Average Pain Intensity (Over a Twelve-week Period)
Description: The participant scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
  Average pain intensity score is the average of pain experienced for previous 24 hours as rated on an 11-point NRS at each visit. Calculations are based on 3 consecutive planned (at 4-weekly intervals) visits.
  All available data of a participant was used; if a participant dropped-out or had incomplete data during a 12-week period no imputations were performed for the missing values.
Time Frame: Day 1; up to Week 144
Population: Safety Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
units on a scale
  Baseline | 3.3 (1.79)
  Week 1 to 12: number analyzed (Participants) | 30
  Week 1 to 12 | 3.1 (1.95)
  Week 13 to 24: number analyzed (Participants) | 20
  Week 13 to 24 | 3.1 (2.51)
  Week 25 to 36: number analyzed (Participants) | 14
  Week 25 to 36 | 2.1 (1.57)
  Week 37 to 48: number analyzed (Participants) | 13
  Week 37 to 48 | 2.0 (1.71)
  Week 49 to 60: number analyzed (Participants) | 11
  Week 49 to 60 | 2.0 (1.78)
  Week 61 to 72: number analyzed (Participants) | 9
  Week 61 to 72 | 2.0 (1.61)
  Week 73 to 84: number analyzed (Participants) | 8
  Week 73 to 84 | 2.4 (1.97)
  Week 85 to 96: number analyzed (Participants) | 7
  Week 85 to 96 | 3.1 (3.16)
  Week 97 to 108: number analyzed (Participants) | 6
  Week 97 to 108 | 3.1 (3.76)
  Week 109 to 120: number analyzed (Participants) | 3
  Week 109 to 120 | 3.3 (2.52)
  Week 121 to 132: number analyzed (Participants) | 1
  Week 121 to 132 | 1.0 (0)
  Week 133 to 144: number analyzed (Participants) | 1
  Week 133 to 144 | 1.0 (0)

6. Other Pre Specified Outcome: Average Daily Total Tapentadol Prolonged Release Dose
Description: The Total Daily Dose (TDD) on any given day is the sum of the morning and evening intake amounts. The average TDD is an individuals average over the trial period.
Time Frame: Day 1; up to 144 weeks
Population: Safety Set.
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
mg per day | 360 (91.21)

7. Secondary Outcome: Tapentadol Prolonged Release Exposure
Description: The number of days that participants took tapentadol prolonged release. The extent of exposure was categorized into 2 periods, less than 90 days and more than 90 days (up to 144 weeks).
Time Frame: Day 1; up to 144 weeks
Population: Safety Set.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 31
participants
  0 to 90 days | 11
  more than 90 days | 20

8. Primary Outcome: Time Dependence of Adverse Events
Description: The onset and duration of TEAEs was not evaluated for this trial.
Time Frame: Day 1; 144 weeks
Population: No evaluation was performed.
Groups:
- Frequency of Treatment Emergent Adverse Events: All participants from the KF5503/15 that enrolled into this trial were on tapentadol prolonged release. Participants were dosed in the range of 100 to 250 mg tapentadol twice daily. The dose was titrated to achieve sufficient pain relief to continue with effective analgesia for as long as the participant tolerated and wishes to continue treatment.
Arm/Group | Frequency of Treatment Emergent Adverse Events
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: One participant was treated up to 144 weeks.
Arm/Group | Tapentadol Prolonged Release
Serious Adverse Events (participants affected / at risk) | 14/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Prolonged Release (N=31)
hypoalbuminaemia (Metabolism and nutrition disorders) | 1 — Treatment emergent event leading to death
azotaemia (Renal and urinary disorders) | 1 — Treatment emergent event leading to death
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 — Investigator indicated that the progression of the underlying malignancy (lung carcinoma) was associated with the hypoxia. Treatment emergent event leading to death.
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 — Treatment emergent event leading to death
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Treatment emergent event leading to death
metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
anaemia (Blood and lymphatic system disorders) | 1
cholecystitis (Hepatobiliary disorders) | 1
pneumonia (Infections and infestations) | 1
cardiac failure (Cardiac disorders) | 1 — Post-treatment adverse event leading to death 30 days after the last administration of tapentadol PR. The participant did not have another serious adverse event.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Prolonged Release (N=31)
Anaemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
nausea (Gastrointestinal disorders) | 9
constipation (Gastrointestinal disorders) | 4
abdominal pain upper (Gastrointestinal disorders) | 2
pyrexia (General disorders) | 4
ascites (Gastrointestinal disorders) | 2
general physical health deterioration (General disorders) | 3
fatigue (General disorders) | 2
dizziness (Nervous system disorders) | 3
headache (Nervous system disorders) | 3
somnolence (Nervous system disorders) | 2
sinus tachycardia (Cardiac disorders) | 3
tachycardia (Cardiac disorders) | 3
bronchitis (Infections and infestations) | 2
urinary tract infection (Infections and infestations) | 2
pathological fracture (Musculoskeletal and connective tissue disorders) | 2
haematuria (Renal and urinary disorders) | 2

LIMITATIONS AND CAVEATS:
The trial was stopped for administrative reasons. Three years after trial initiation 2 participants were in the trial and to permit analysis and reporting the sponsor decided to terminate the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.